CLINICAL TRIAL: NCT03577990
Title: An Interactive Technology Enhanced Coaching Intervention for Black Women With Hypertension
Brief Title: Technology Coaching Intervention for Black Women With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Charlotte (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Willie Abel, Assistant Professor, University of North Carolina, Charlotte
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0549; 1K01HL140288 (NIH)
Record Dates: First submitted 2018-04-18; First posted 2018-07-05 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-04

CONDITIONS: Uncontrolled Hypertension
Keywords: hypertension, Black women, self-management, coaching
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The study will test the effects of ITEC added to CDSMP on two study aims: 1) BP control, and 2) adherence to antihypertensive medication and lifestyle modifications. After baseline data collection, participants complete a 6-week CDSMP course and then are randomly assigned to either the treatment or control arm. All participants will continue to receive usual care for HTN.
  The treatment group will receive ITEC and wireless tools to track activity, BP, weight, food intake, and self-report medication-taking after an orientation to Fitbit Plus (a cloud-based collaborative care platform designed to store and track data). All tools will be synced to the participants' smartphone. The treatment arm will receive weekly ITEC for 3 months, biweekly ITEC for 3 months, and then no ITEC for 3 months.
  The control arm will receive usual care only with monthly BP measured manually for 3 months and then receive the same wireless tools with monitoring to track comparative data with the treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Technology Enhanced Coaching (ITEC) (Experimental): Fitbit Plus monitoring will include BP, weight measurements, daily food intake, self-report medication-taking, and physical activity plus weekly Interactive Technology-Enhanced Coaching (ITEC) for 3 months, then biweekly ITEC for 3 months, followed by another 3 months with no coaching to assess for sustainability.
  Interventions: Behavioral: Interactive Technology Enhanced Coaching (ITEC)
- Interactive Technology-No Coaching (IT) (Active Comparator): Participants will receive usual care for 3 months followed by 6 months of only Fitbit Plus monitoring (with no ITEC) of BP, weight measurements, daily food intake, self-report medication-taking, and physical activity to be used for comparative data with the treatment arm.
  Interventions: Behavioral: Interactive Technology-No Coaching (IT)

INTERVENTIONS:
Behavioral: Interactive Technology Enhanced Coaching (ITEC) — As participants wear the activity tracker, take their BP and weight, along with input of food intake and medication-taking, data is transmitted in real time via Bluetooth Smart technology to the Fitbit Plus dashboard. All data is tracked, analyzed, and transparently displayed for participants to view and better understand their condition, and actively engage in self-care. Staff monitor data and communicate with participants to encourage active engagement in action plans by sending tailored coaching messages (ITEC) via the Fitbit Plus dashboard to the treatment arm weekly for 3 months, and biweekly for 3 months to motivate and support (BP control, medication adherence, and lifestyle modifications). After 6 months, the treatment arm will be monitored an additional 3 months with no tailored coaching for sustainability.
  Arms: Interactive Technology Enhanced Coaching (ITEC)
Behavioral: Interactive Technology-No Coaching (IT) — After receiving usual care for 3 months, the control arm will receive the same electronic monitoring as the treatment arm and data will be captured in the same manner with the Fitbit Plus dashboard. Participants will be expected to use the information from the dashboard and the CDSMP workshop as a guide to self-care without coaching (IT). Staff will only monitor data. Control participants will not be contacted between repeated measures data collection periods, except to send reminders if they are not participating daily.
  Arms: Interactive Technology-No Coaching (IT)

SUMMARY:
Hypertension (HTN) is a global problem affecting 972 million adults and an important public health burden since it is the main cause of cardiovascular disease and death, and the second leading cause of disability. Disproportionately affected, Black women have the highest prevalence of HTN in the United States. This research will evaluate potential interventions for possible community-based strategies for controlling HTN using interactive self-care strategies with coaching and technology. We hypothesize that participants who receive the Chronic Disease Self-Management Program (CDSMP) workshop and Interactive Technology Enhanced Coaching (ITEC) will have lower systolic/diastolic blood pressure (BP) and better adherence to antihypertensive medication(s) and lifestyle recommendations (physical activity, diet, and weight management) post intervention compared to participants receiving self-care management alone.

DETAILED DESCRIPTION:
This study includes a sample of community dwelling Black women with uncontrolled HTN. All participants meeting study eligibility requirements will receive the Chronic Disease Self-Management Program (CDSMP) workshop for 6 weeks. Participants from this pool will be randomized to the treatment and control arm. All study participants will continue to receive usual care for their HTN.

The intervention will be divided into three steps. At Step 1 for 3 months, the treatment arm will receive electronic monitoring (of participants' BP, weight, physical activity, food diary, and medication-taking) with weekly Interactive Technology Enhanced Coaching (ITEC) while the control arm will receive usual care with manual BP measurements monthly. At Step 2 for three months, the treatment arm will receive electronic monitoring with ITEC biweekly, and the control arm will receive electronic monitoring only. At Step 3 for three months, both the treatment arm and the control arm will receive electronic monitoring only.

Our sample of n=45 participants per arm (N=90 in total), will be measured (electronic measurements, anthropometric measurements, and data collection tools) at baseline, 3 months, 6 months, and at 9 months post CDSMP. A hierarchical, mixed-effects repeated measures design will be used to analyze the data.

The project is a two-arm randomized controlled trial with specific aims to determine whether the effects of CDSMP combined with ITEC will maintain BP control, attain medication adherence, and achieve lifestyle modifications (physical activity, diet, and weight management) compared to the CDSMP alone. We will test the hypothesis that:

1. More participants in the CDSMP/ITEC arm will have controlled BP less than 130/80 at 3 months, 6 months, and at 9 months post CDSMP, compared to participants in CDSMP alone.
2. More participants in the CDSMP/ITEC arm will have higher levels of adherence to antihypertensive medication(s) at 3 months, 6 months, and at 9 months post CDSMP, compared to participants in the CDSMP alone.
3. More participants in the CDSMP/ITEC arm, will have higher levels of adherence to lifestyle modifications (physical activity, diet, and weight management) at 3 months, 6 months, and at 9 months post CDSMP, compared to participants in the CDSMP alone.

Information from this study may be used to enhance self-care management, control blood pressure, and increase the quality of life for Black women who are burdened with the adverse effects of HTN and its high disability and mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as Black or African American;
* 18-70 years of age
* English speaking
* Has to live in the study community, Charlotte or surrounding area
* Systolic BP greater than or equal to 130 and/or diastolic BP greater than or equal to 80 at screening
* Prescribed to take one or more antihypertensive medication(s)
* Smartphone or device
* Bluetooth 4.0 and Provider network or Wi-Fi connectivity

Exclusion Criteria:

* Self-report of mental illness that interferes with daily functioning
* Unable to be physically active
* Current pregnancy
* Plans to move from the study area during the project
* Systolic BP greater than or equal to 160 and/or diastolic BP greater than or equal to 100
* Uncontrolled diabetes (HbA1c >8.5), hemodialysis, stroke (within past year with residual effects such as weakness, paralysis, speech difficulty, etc.), cancer treatment (for spread of cancer to other places in the body), or a heart attack (within the past year)
* Concurrent participation in another research study and/or taken any Stanford self-management program

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willie M Abel, PhD, Principal Investigator — The University of North Carolina at Charlotte; Mark J DeHaven, PhD, Study Director — The University of North Carolina at Charlotte
Locations (1):
- Churches, Salons, Community Events, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abel WM, Spikes T, Greer DB. A Qualitative Study: Hypertension Stigma Among Black Women: Erratum. J Cardiovasc Nurs. 2025 May-Jun 01;40(3):279. doi: 10.1097/JCN.0000000000001213. No abstract available. PMID 40198262
- [Derived] Abel WM, DeHaven MJ. An interactive technology enhanced coaching intervention for Black women with hypertension: Randomized controlled trial study protocol. Res Nurs Health. 2021 Feb;44(1):24-36. doi: 10.1002/nur.22090. Epub 2020 Dec 15. PMID 33319386

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from areas frequented by Black women, including churches, sororities, clubs, community associations, neighborhood schools, and community events between January 2019 and April 2019. The first participant was enrolled on January 28, 2019, and the last participant was enrolled on April 13, 2019.
Pre-assignment Details: Of the 166 individuals approached for enrollment, 40 did not meet the inclusion criteria, 36 declined to participate, while 90 met the inclusion criteria and consented to participate in the study. The 90 participants were enrolled in the 6-week Chronic Disease Self-Management Program (CDSMP), and 83 completed the program and were randomized to treatment. Of the 83 participants, 77 had Fitbit data for analysis.
Groups:
- Interactive Technology Enhanced Coaching (ITEC): Fitbit Plus monitoring will include BP, weight measurements, daily food intake, self-report medication-taking, and physical activity plus weekly Interactive Technology-Enhanced Coaching (ITEC) for 3 months, then biweekly ITEC for 3 months, followed by another 3 months with no coaching to assess for sustainability.
  Interactive Technology Enhanced Coaching (ITEC): As participants wear the activity tracker, take their BP and weight, along with input of food intake and medication-taking, data is transmitted in real time via Bluetooth Smart technology to the Fitbit Plus dashboard. All data is tracked, analyzed, and transparently displayed for participants to view and better understand their condition, and actively engage in self-care. Participants will be expected to use the information from the Fitbit dashboard and the Chronic Disease Self-Management Program (CDSMP) workshop as a guide to self-care. In addition, staff will monitor data and communicate with participants to encourage active engagement in action plans by sending tailored coaching messages (ITEC) via the Fitbit Plus dashboard to the treatment arm weekly for 3 months, and biweekly for 3 months to motivate and support (BP control, medication adherence, and lifestyle modifications). After 6 months, the treatment arm will be monitored an additional 3 months with no tailored coaching for sustainability.
  Data were collected and compared at 3, 6, and 9 months.
- Interactive Technology-No Coaching (IT): Participants will receive usual care for 3 months followed by 6 months of only Fitbit Plus monitoring (with no ITEC) of BP, weight measurements, daily food intake, self-report medication-taking, and physical activity to be used for comparative data with the treatment arm.
  Interactive Technology-No Coaching (IT): After receiving usual care for 3 months, the control arm will receive the same electronic monitoring as the treatment arm and data will be captured in the same manner with the Fitbit Plus dashboard. Participants will be expected to use the information from the dashboard and the Chronic Disease Self-Management Program (CDSMP) workshop as a guide to self-care without coaching (IT). Staff will only monitor data. Control participants will not be contacted between repeated measures data collection periods, except to send reminders if they are not participating daily.
  Data were collected and compared at 3, 6, and 9 months.
Period: Overall Study
Arm/Group | Interactive Technology Enhanced Coaching (ITEC) | Interactive Technology-No Coaching (IT)
Started | 45 | 45
Month 1-3 | 42 | 41
Month 4-6 | 41 | 39
Month 7-9 | 38 | 34
Completed | 37 | 32
Not Completed | 8 | 13
Not completed — Lost to Follow-up | 4 | 6
Not completed — Withdrawal by Subject | 4 | 7

BASELINE CHARACTERISTICS:
Population: 90 participants were enrolled in the 6-week Chronic Disease Self-Management Program (CDSMP), and 83 completed the program and were randomized to treatment.
Groups:
- Interactive Technology Enhanced Coaching (ITEC): Chronic Disease Self-Management Program (CDSMP) and interactive technology using the smartphone for self-monitoring of 1) blood pressure with the Omron 10 wireless Bluetooth home BP monitor (Model BP786N), 2) medication adherence by checking each time medication was taken within the Fitbit Platform, 3) daily steps with the Fitbit Inspire HR activity tracker, 4) food intake (calories and sodium) with MyFitnessPal, and 5) weight with Fitbit Aria 2 weight scale, along with coaching by means of personalized text messages.
  Data were collected and compared at 3, 6, and 9 months.
- Interactive Technology-No Coaching (IT): Chronic Disease Self-Management Program (CDSMP) and interactive technology using the smartphone for self-monitoring of 1) blood pressure with the Omron 10 wireless Bluetooth home BP monitor (Model BP786N), 2) medication adherence by checking each time medication was taken within the Fitbit Platform, 3) daily steps with the Fitbit Inspire HR activity tracker, 4) food intake (calories and sodium) with MyFitnessPal, and 5) weight with Fitbit Aria 2 weight scale.
  Data were collected and compared at 3, 6, and 9 months.
- Total: Total of all reporting groups
Arm/Group | Interactive Technology Enhanced Coaching (ITEC) | Interactive Technology-No Coaching (IT) | Total
Number analyzed (Participants) | 42 | 41 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 36 | 35 | 71
  >=65 years | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (8.6) | 52.7 (11.0) | 54.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 83
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 41 | 83
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 41 | 83
Years with Hypertension [Mean (Standard Deviation); unit: years] | 11.0 (8.1) | 9.8 (8.0) | 10.4 (8.0)
Marital Status [Count of Participants; unit: Participants]
  Single (never married) | 10 | 12 | 22
  Married | 18 | 18 | 36
  Separated/Divorced | 12 | 9 | 21
  Widowed | 2 | 2 | 4
Education [Count of Participants; unit: Participants]
  Less than 12th grade | 0 | 1 | 1
  Completed high school | 0 | 2 | 2
  Some community college | 7 | 4 | 11
  Completed community college | 3 | 4 | 7
  Some 4-year college | 3 | 5 | 8
  Completed 4-year college | 18 | 10 | 28
  Some graduate school | 1 | 1 | 2
  Completed graduate school | 10 | 14 | 24
Income [Count of Participants; unit: Participants]
  <10,000 - 24,999 | 6 | 5 | 11
  25,000 - 54,999 | 14 | 12 | 26
  55,000 - >100,000 | 21 | 23 | 44
  Refused | 1 | 1 | 2
Occupational Status [Count of Participants; unit: Participants]
  Work full-time | 27 | 33 | 60
  Work part-time / Not employed | 7 | 3 | 10
  Retired with pension | 8 | 5 | 13
Baseline systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 140.1 (11.0) | 139.0 (9.0) | 139.6 (10.0)
Baseline diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 83.9 (8.6) | 84.3 (7.0) | 84.1 (7.8)
Baseline weight [Mean (Standard Deviation); unit: pounds] | 213.5 (47.2) | 214.3 (52.2) | 213.9 (49.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic and Diastolic Blood Pressure (BP)
Description: To show the change (decrease) in systolic blood pressure (SBP) and diastolic blood pressure (DBP) over 9 months.
Time Frame: Baseline to 3 months, 6 months, and 9 months.
Population: Numbers may have decreased over time due to attrition and/or non-participation.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Interactive Technology Enhanced Coaching (ITEC) | Interactive Technology-No Coaching (IT)
Number analyzed (Participants) | 42 | 41
mmHg
  Baseline Systolic BP | 140.07 (1.5781) | 139.03 (1.6841)
  Month 3 Systolic BP: number analyzed (Participants) | 41 | 36
  Month 3 Systolic BP | 124.18 (1.9429) | 128.31 (1.9737)
  Month 6 Systolic BP: number analyzed (Participants) | 41 | 36
  Month 6 Systolic BP | 125.80 (1.9606) | 126.13 (2.0827)
  Month 9 Systolic BP: number analyzed (Participants) | 41 | 36
  Month 9 Systolic BP | 125.04 (1.7349) | 125.67 (1.8618)
  Baseline Diastolic BP: number analyzed (Participants) | 41 | 36
  Baseline Diastolic BP | 83.8578 (1.2306) | 84.3161 (1.3132)
  Month 3 Diastolic BP: number analyzed (Participants) | 41 | 36
  Month 3 Diastolic BP | 82.8319 (1.4629) | 79.9767 (1.4749)
  Month 6 Diastolic BP: number analyzed (Participants) | 41 | 36
  Month 6 Diastolic BP | 83.2099 (1.3628) | 82.3126 (1.4482)
  Month 9 Diastolic BP: number analyzed (Participants) | 41 | 36
  Month 9 Diastolic BP | 82.5838 (1.4368) | 81.6017 (1.5639)

2. Secondary Outcome: Medication Adherence by Proportion of Days Covered
Description: To show the proportion of days covered in the period of interest (Month 1, Month 3, Month 6, and Month 9). (Sum of days covered that participant reported medication adherence in the period of interest) ÷ (the number of days in the period of interest) x 100.
Time Frame: Month 1 to Month 3, Month 6, and Month 9.
Population: In the IT arm, months 1-3, participants received usual care with no data collection and thus, there are no entries in these rows on the table. The information provided in the 'Other Statistical Analysis' field below clarifies that for the IT arm, months 1-6 in the statistical analysis corresponds to calendar months 4-9 of the data collection.
Measure: Least Squares Mean (Standard Error); unit: Proportion of days
Groups:
- Interactive Technology-No Coaching (IT): Participants will receive usual care for 3 months (with no Fitbit monitoring data collected) followed by 6 months of only Fitbit Plus monitoring (with no ITEC) of BP, weight measurements, daily food intake, self-report medication-taking, and physical activity to be used for comparative data with the treatment arm.
  Interactive Technology-No Coaching (IT): After receiving usual care for 3 months, the control arm will receive the same electronic monitoring as the treatment arm and data will be captured in the same manner with the Fitbit Plus dashboard. Participants will be expected to use the information from the dashboard and the Chronic Disease Self-Management Program (CDSMP) workshop as a guide to self-care without coaching (IT). Staff will only monitor data. Control participants will not be contacted between repeated measures data collection periods, except to send reminders if they are not participating daily.
  Data were collected and compared at 3, 6, and 9 months.
Arm/Group | Interactive Technology Enhanced Coaching (ITEC) | Interactive Technology-No Coaching (IT)
Number analyzed (Participants) | 41 | 36
Proportion of days
  Month 1 Med Adherence: number analyzed (Participants) | 41 | 0
  Month 1 Med Adherence | 0.7404 (0.06353) |
  Month 3 Med Adherence: number analyzed (Participants) | 41 | 0
  Month 3 Med Adherence | 0.6507 (0.06353) |
  Month 6 Med Adherence | 0.5575 (0.06353) | 0.5357 (0.06779)
  Month 9 Med Adherence | 0.6507 (0.06353) | 0.5595 (0.06779)
Statistical Analysis 1: Comparison: Interactive Technology Enhanced Coaching (ITEC) vs Interactive Technology-No Coaching (IT); Test type: Superiority — Our sample (N = 90) had approximately 80% power (assuming 5 dropouts per arm) to detect an effect size of ∼.205 or greater at the α = .05 level of statistical significance, given a realistic range of simulated unstructured covariance matrices. An 11% rate of attrition was anticipated to yield a final sample of 80 participants, an average of 40 per arm. Participants who dropped out of the study prior to receiving the allotted intervention were not included in the analysis; p = .05, mixed-effects repeated measures — P-values were computed according to a mixed-effects repeated measures model, appropriately constrained to baseline if indicated; Mean Difference (Final Values) = .125; For both referent (compared by month and treatment group) and constrained longitudinal data analysis (cLDA) models, p-values were computed for the main group (G), time (T), and interaction (G x T) effects. For the first 3 months of the referent arm (IT), data were compared with usual care. Consequently, months 1 - 6 in the statistical analysis corresponds to calendar months 4 - 9 of the data collection. Months 1 - 9 of the intervention arm (ITEC) reflects months 1 - 9 of the collection. Additionally, for the cLDA model, data in the referent arm (IT) were accordingly shifted such that the starting point on the y-axis for both arms were the same (i.e. y = 0)

3. Secondary Outcome: Physical Activity (Change in Daily Steps)
Description: To show the change (increase) in daily steps over 9 months.
Time Frame: Month 1 to Month 3, Month 6, and Month 9.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: steps
Arm/Group | Interactive Technology Enhanced Coaching (ITEC) | Interactive Technology-No Coaching (IT)
Number analyzed (Participants) | 41 | 34
steps
  Month 1 Steps: number analyzed (Participants) | 41 | 0
  Month 1 Steps | 5778.58 (555.38) |
  Month 3 Steps: number analyzed (Participants) | 41 | 0
  Month 3 Steps | 5384.34 (593.17) |
  Month 6 Steps | 4720.90 (611.08) | 6413.73 (663.43)
  Month 9 Steps | 4743.20 (770.29) | 5092.30 (798.81)
Statistical Analysis 1: Comparison: Interactive Technology Enhanced Coaching (ITEC) vs Interactive Technology-No Coaching (IT); Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .05, mixed-effects repeated measures — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1250; [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: Change in Dietary Intake (Calories)
Description: To show the change (decrease) in dietary intake (calories) over 9 months.
Time Frame: Month 1 to Month 3, Month 6, and Month 9.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: calories
Arm/Group | Interactive Technology Enhanced Coaching (ITEC) | Interactive Technology-No Coaching (IT)
Number analyzed (Participants) | 41 | 30
calories
  Month 1 Calories: number analyzed (Participants) | 41 | 0
  Month 1 Calories | 1204.75 (81.7083) |
  Month 3 Calories: number analyzed (Participants) | 41 | 0
  Month 3 Calories | 1133.66 (92.0513) |
  Month 6 Calories | 801.42 (96.8770) | 803.38 (122.88)
  Month 9 Calories | 1247.33 (146.01) | 1029.74 (165.78)
Statistical Analysis 1: Comparison: Interactive Technology Enhanced Coaching (ITEC) vs Interactive Technology-No Coaching (IT); Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .05, mixed-effects repeated measures — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 300; [other analysis details as in outcome 2, analysis 1]

5. Secondary Outcome: Change in Weight
Description: To show the change (decrease) in weight over 9 months.
Time Frame: Baseline to 3 months, 6 months, and 9 months.
Population: Numbers may have decreased over time due to attrition and/or non-participation.
Measure: Least Squares Mean (Standard Error); unit: pounds
Arm/Group | Interactive Technology Enhanced Coaching (ITEC) | Interactive Technology-No Coaching (IT)
Number analyzed (Participants) | 42 | 41
pounds
  Baseline Weight | 213.54 (7.6390) | 214.31 (8.1523)
  Month 3 Weight: number analyzed (Participants) | 41 | 36
  Month 3 Weight | 205.23 (7.6767) | 212.20 (8.1523)
  Month 6 Weight: number analyzed (Participants) | 41 | 36
  Month 6 Weight | 203.71 (7.7075) | 203.71 (8.2126)
  Month 9 Weight: number analyzed (Participants) | 41 | 36
  Month 9 Weight | 202.36 (7.8919) | 205.40 (8.4171)

6. Secondary Outcome: Change in Dietary Intake (Sodium)
Description: To show the change (decrease) in dietary intake (sodium) over 9 months.
Time Frame: Month 1 to Month 3, Month 6, and Month 9.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | Interactive Technology Enhanced Coaching (ITEC) | Interactive Technology-No Coaching (IT)
Number analyzed (Participants) | 41 | 30
mg
  Month 1 Sodium: number analyzed (Participants) | 41 | 0
  Month 1 Sodium | 1363.65 (116.66) |
  Month 3 Sodium: number analyzed (Participants) | 41 | 0
  Month 3 Sodium | 1386.61 (134.26) |
  Month 6 Sodium | 775.66 (141.33) | 928.30 (181.33)
  Month 9 Sodium | 1226.89 (179.26) | 1512.05 (241.61)
Statistical Analysis 1: Comparison: Interactive Technology Enhanced Coaching (ITEC) vs Interactive Technology-No Coaching (IT); Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = .05, mixed-effects repeated measures — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 500; [other analysis details as in outcome 2, analysis 1]

7. Other Pre Specified Outcome: Stigma and Hypertension, Qualitative Study
Description: Qualitative questionnaire (included written responses to two open-ended questions) to gain insight and describe the psychological factor of stigma as an influence on poorly controlled hypertension in Black women. No scale was used to assess data.
Time Frame: 15 minutes
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 42 weeks. Includes 6-week Chronic Disease Self-Management Program and 36 weeks of data collection.
Description: Definitions do not differ.
Arm/Group | Interactive Technology Enhanced Coaching (ITEC) | Interactive Technology-No Coaching (IT)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 9/42 | 3/41
Other Adverse Events (participants affected / at risk) | 0/42 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interactive Technology Enhanced Coaching (ITEC) (N=42) | Interactive Technology-No Coaching (IT) (N=41)
Stroke (Vascular disorders) | 0 (0) | 1 (1) — Hospitalized with stroke following colonoscopy procedure. Withdrew from study.
Elevated diastolic blood pressure >110 (Vascular disorders) | 1 (1) | 0 (0) — Hospitalized with diastolic blood pressure >110. Anti-hypertensive medications re-evaluated and diastolic blood pressure decreased gradually to 90s.
Dislodged patella (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Dislodged patella left knee - old injury. Participant minimized this pre-existing condition when assessing for study eligibility. Outpatient treatment, may require surgery.
Twisted ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Twisted ankle and damaged Achilles from fall at work. Treated as outpatient. Recovered without incident.
Bunion surgery (Surgical and medical procedures) | 1 (1) | 0 (0) — Elective Bunion surgery. Participant minimized pre-existing condition when assessing for study eligibility. Uneventful recovery.
Total knee replacement (Surgical and medical procedures) | 1 (1) | 0 (0) — Surgery and hospitalization for total knee replacement due to increased pain. Participant minimized pre-existing condition when assessing for study eligibility. Follow-up with outpatient rehabilitation. Uneventful recovery.
Shoulder replacement (Surgical and medical procedures) | 1 (1) | 0 (0) — Surgery and hospitalization for shoulder replacement due to increased pain. Participant minimized pre-existing condition when assessing for study eligibility. Follow-up with outpatient rehabilitation. Uneventful recovery.
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Breast cancer returned after remission with metastasis. Withdrew from study.
Glaucoma (Surgical and medical procedures) | 1 (1) | 0 (0) — Outpatient surgery for glaucoma. Participant did not mention this pre-existing condition when assessing for study eligibility. Recovered without incident.
Abdominal pain and bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) — Hospitalized for abdominal pain and bleeding. Recovered without incident.
Stomach virus (Gastrointestinal disorders) | 1 (1) | 0 (0) — Hospitalized for stomach virus. Recovered without incident.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Treated as an outpatient for pneumonia. Recovered without incident.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT03577990/Prot_SAP_000.pdf